CLINICAL TRIAL: NCT00053638
Title: A Phase III, Randomized, Open-label, Multicenter Study of the Safety and Efficacy of Efavirenz Versus Tenofovir When Administered in Combination With the Abacavir/Lamivudine Fixed-dose Combination Tablet as a Once-daily Regimen in Antiretroviral-naive HIV-1 Infected Subjects.
Brief Title: A New Tablet Containing Two FDA-Approved Drugs In HIV-Infected Patients Who Have Not Received Prior Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESS30009
Record Dates: First submitted 2003-02-04; First posted 2003-02-05 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infection
Keywords: HIV-1 Efavirenz Tenofovir
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Tenofovir; abacavir, lamivudine drug combination

INTERVENTIONS:
Drug: efavirenz
Drug: tenofovir
Drug: abacavir/lamivudine
  Other Names: efavirenz; tenofovir

SUMMARY:
This is a 48-week study to evaluate the safety and efficacy of a new tablet formulation containing two FDA-approved drugs in HIV-infected patients who have not received prior therapy. This tablet will be taken with one of two FDA-approved drugs as a once-daily regimen. Study physicians will evaluate subjects to determine if they have certain medical conditions, laboratory test values, medication use, or drug allergies that would exclude them from the study.

ELIGIBILITY:
Inclusion criteria:

* Participants must be able to provide informed consent.
* Have documented HIV-1 infection.
* Have not received more than 14 days of prior treatment with antiretroviral drugs.
* Meet laboratory test criteria.
* Women of childbearing potential must abstain from sexual intercourse or use acceptable contraception.
* Must be able to take study medications as directed and complete all study visits and evaluations during the 48 week study.

Exclusion criteria:

* Enrolled in other HIV treatment studies.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345
Dates: Start 2003-02; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Viral load response at 48 weeks | 48 weeks

SECONDARY OUTCOMES:
Safety and tolerability Viral load response at 24 weeks Change in T-cell count Resistance Pharmacokinetics | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (45):
- United States (45):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Reading, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Green Bay, Wisconsin

REFERENCES:
- [Derived] Underwood MR, Ross LL, Irlbeck DM, Gerondelis P, Rouse E, St Clair MH, Trinh L, Parkin N, Lanier E. Sensitivity of phenotypic susceptibility analyses for nonthymidine nucleoside analogues conferred by K65R or M184V in mixtures with wild-type HIV-1. J Infect Dis. 2009 Jan 1;199(1):84-8. doi: 10.1086/595296. PMID 19032103